CLINICAL TRIAL: NCT01909765
Title: Comparison of Two Different Circumcision Surgical Technique on Postoperative Pain
Brief Title: Two Different Surgical Techniques on Postoperative Circumcision Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Reyhan Polat, Medical Doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: Circumcicsion
Record Dates: First submitted 2013-07-18; First posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Postoperative Pain
Keywords: Circumcision; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Wound Closure Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dorsal slite (Active Comparator): Skin and mucosa insicion made together
  Interventions: Other: Dorsal slit
- Double incision (Experimental): Skin and mucosa incision made separately
  Interventions: Other: Double incision

INTERVENTIONS:
Other: Dorsal slit — Skin and mucosa incision made together
  Arms: Dorsal slite
Other: Double incision — Skin and mucosa incision made separately
  Other Names: Surgical technique
  Arms: Double incision

SUMMARY:
To compare the effect of two different surgical techniques, the dorsal slit and double incision technique, on postoperative pain.

DETAILED DESCRIPTION:
Two different circumcision techniques result in different kinds of pain.This research aims determine which is more beneficial to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Children

Exclusion Criteria:

* Patients with any bleeding

Ages: 2 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
To asses postoperative pain scores on Modified Objective Assessment Scale (MOAS) | Postoperative first two hours

CONTACTS AND LOCATIONS:
Overall Officials: Reyhan Polat, MD, Principal Investigator — Yildirim Beyazit Education and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Education and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Karakoyunlu N, Polat R, Aydin GB, Ergil J, Akkaya T, Ersoy H. Effect of two surgical circumcision procedures on postoperative pain: A prospective, randomized, double-blind study. J Pediatr Urol. 2015 Jun;11(3):124.e1-5. doi: 10.1016/j.jpurol.2015.01.002. Epub 2015 Mar 3. PMID 25842991